CLINICAL TRIAL: NCT06538974
Title: Adherence to Long-term Exoskeleton Rehabilitation to Treat Lower Limb Weakness and / or Deficiencies in Adult Population
Acronym: ALERT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wandercraft (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP005 ALERT
Record Dates: First submitted 2024-07-09; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Motor Disorders; Gait Disorders, Neurologic; Neurodegenerative Diseases; Spinal Cord Injuries; Weakness, Muscle; Cerebrovascular Accident
Keywords: Hands-free Exoskeleton; Atalante X; Gait; Balance; Rehabilitation
MeSH Terms: conditions — Motor Disorders; Gait Disorders, Neurologic; Neurodegenerative Diseases; Spinal Cord Injuries; Muscle Weakness; Stroke

STUDY DESIGN:
Intervention Model Description: Adult patients presenting lower limb weakness and / or deficiencies, regardless of the underlying causes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hands-free exoskeleton (Experimental)
  Interventions: Device: Hands-free exoskeleton

INTERVENTIONS:
Device: Hands-free exoskeleton — During the one-year intervention period, participants will complete at least one exoskeleton session per week (≥36 sessions) with the Atalante X. The additional voluntary year follows the same design. During sessions with the exoskeleton, the patients will perform ambulatory exercises with the device, with a gradual increase of intensity through the sessions.

SUMMARY:
In 2019, approximately 2.4 billion people worldwide required rehabilitation for various health pathologies, a 63% increase since 1990. It has been suggested that current rehabilitation frameworks (inpatient, outpatient, and community-based) are insufficient to meet local population needs due to issues like long waiting times, lack of facilities, prioritization, funding, and accessibility.Patients with lower limb weaknesses, resulting from various conditions (for example stroke, traumatic brain injury, spinal cord injury and others) require long-term management and motivation for engagement, which are crucial for functional outcomes. This highlights the need for sustainable gait and balance rehabilitation.

New technologies like exoskeletons have shown promising results in short-term inpatient programs, improving gait, balance, and quality of life, however, long-term follow-up data are still needed.

The present clinical investigation is a national, prospective, open-label interventional trial, proposing a 12-month outpatient rehabilitation program with the Atalante X exoskeleton to treat lower limb weakness and/or impairments in 100 participants. The rehabilitation program consists of at least one exoskeleton rehabilitation session per week. At the end of the first-year experimental phase, participants can continue for an additional year in the voluntary phase. The program aims to explore the potential long-term effects of supervised robotic rehabilitation on motor, cognitive, bowel, bladder functions, quality of life, and well-being. Assessments are conducted at baseline, after 4 and 12 months of exoskeleton rehabilitation, and at 16 and 24 months for participants in the voluntary phase.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from lower limb weaknesses and / or deficiencies regardless of the cause
* Adult patient ≥18 years old
* Patient able to read and write in French and who have signed an informed consent form
* Patient affiliated to a social security system.

Exclusion Criteria:

* Individual with severe spasticity of adductor muscles, hamstring, quadriceps and triceps surae. Severe spasticity is defined by a score of 4 on the modified Ashworth scale
* Pregnant woman
* Individual with history of osteoporotic fracture and / or pathology or treatment causing secondary osteoporosis
* Pressure Ulcer of Grade I or higher according to the NPUAP International Pressure Ulcer Classification System- EPUAP, in areas of contact with the Atalante X system
* Severe aphasia limiting ability to express needs or to fulfil questionnaires, at the discretion of the physician.
* Patient with a cardiac or respiratory contraindication to physical exertion, at discretion of the physician
* Patient unable to deliver his/her consent
* Patient under legal protection
* Patient participating at the same time in another study
* Patients with morphological contraindications to the use of the Atalante X exoskeleton (as per user's manual) with exceptions as follows: knee flessum of 20° authorized if sensibility is present; equinus of the ankle of 20° allowed regardless of presence or absence of sensibility, hip flessum of 20° allowed regardless of presence or absence of sensibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2027-07-02 (Estimated); Study Completion 2027-07-02 (Estimated)

PRIMARY OUTCOMES:
Function in Sitting Test | At baseline, at 4 and 12 months; at 16 and 24 months
  The Function in Sitting Test consists of 14 items, each scored on a scale from 0 to 4, where 0 indicates the lowest ability and 4 represents normal sitting abilities. The maximum achievable score is 56, reflecting normal ability.

SECONDARY OUTCOMES:
10-meter walk test | At baseline, at 4 and 12 months; at 16 and 24 months
  Gait speed during 10 meter walk
Modified Clinical Test of Sensory Integration in Balance | At baseline, at 4 and 12 months; at 16 and 24 months
  Modified Clinical Test of Sensory Integration in Balance test evaluates how different sensory inputs contribute to balance control by assessing balance tasks performed under different sensory conditions: eyes open, firm surface; eyes closed, firm surface; eyes open, foam surface; and eyes closed, foam surface. Scores are based on the time the participant can maintain balance (0-30 seconds for each task, with the maximum score being 120 seconds for all tasks, higher scores reflecting good sensory integration and balance control).
Timed Up and Go | At baseline, at 4 and 12 months; at 16 and 24 months
  Timed Up and Go is a timed task where patient is asked to stand up from the chair, walk 3 meters, turn around, walk and sit again. Based on established thresholds in the literature for various pathologies, the test helps determine if the participant is at risk of falling.
Functional Independence Measure | At baseline, at 4 and 12 months; at 16 and 24 months
  Functional Independence Measure scale score measures the level of disability and the amount of assistance required for an individual to perform activities of daily living. The total score ranges from 18 to 126, with higher scores indicating greater independence.
6-minute walk test | At baseline, at 4 and 12 months; at 16 and 24 months
  6-minute walk test measures the walked distance during a 6 minutes' walk, thus assessing walking endurance and aerobic capacities. Results are compared to normative values based on population-specific references available in the literature.
A five-step clinical assessment of spasticity | At baseline, at 4 and 12 months; at 16 and 24 months
  A five-step clinical assessment of spasticity is used to assess adductor muscles, gluteus maximus, hamstrings, rectus femoris, gastrocnemius and soleus.
Biering-Sorensen test | At baseline, at 4 and 12 months; at 16 and 24 months
  Biering-Sorensen test measures isometric endurance of the trunk extensor muscles, higher times reflecting better endurance.
Muscle strength | At baseline, at 4 and 12 months, at 16 and 24 months
  Hip flexion, extension, abduction, adduction, knee flexion and extension, plantar flexion and extension muscle strength is assessed by using a dynamometer measure (expressed in Newton).
Montreal Cognitive Assessment | At baseline, at 4 and 12 months; at 16 and 24 months
  Montreal Cognitive Assessment is a cognition assessment with scores ranging from 0 to 30, the latter signifying a normal cognitive function.
Adverse events monitoring | Through study completion, up to 24 months for each participant
  Safety is monitored through adverse events occurrence.
Modified Borg Rating of Perceived Exertion | At baseline, at 4 and 12 months, at 16 and 24 months
  Modified Borg Rating of Perceived Exertion measures a level of perceived effort and exertion, breathlessness and fatigue during physical activity with rating going from 0 - nothing at all to 10 - meaning almost maximal effort.
System Usability Scale | At baseline, at 4 and 12 months; at 16 and 24 months
  System Usability Scale measures usability of the exoskeleton training. The scores are from 0 to 100, scores above 72.5 reflecting good usability.
General satisfaction questionnaire | At baseline, at 4 and 12 months; at 16 and 24 months
  General satisfaction is assessed by 3-item questionnaire, assessing interest, satisfaction and level of discomfort. The score is comprised from 0 to 10, higher scores reflecting higher satisfaction following the assessed exoskeleton session.
Specific acceptability | At baseline, at 4 and 12 months; at 16 and 24 months
  Specific acceptability is assessed by five-item questionnaire evaluating participants feedback on post-session anxiety, motivation, safety, fatigue and pain.The score is comprised from 0 to 10, higher scores reflecting higher perceived specific acceptability following the assessed exoskeleton session.
Medical Outcomes Study Short Form 36 | At baseline, at 4 and 12 months; at 16 and 24 months
  Medical Outcomes Study Short Form 36 (SF-36) assesses health related quality of life, by evaluating 8 subdimensions which concern physical functioning, role physical, bodily pain, general health, vitality, social functioning, emotional, and mental health. Two summary scores can be retrieved from the questionnaire: physical health and mental health. For people unable to walk, thus using wheelchair, additional three questions will be added from SF-36 walk-wheel questionnaire. Each domain is scored separately, and scores range from 0 to 100. The higher scores indicate better health status.
Neurogenic bowel dysfunction score | At baseline, at 4 and 12 months; at 16 and 24 months
  Neurogenic bowel dysfunction score measures bowel function, having the scores ranging from 0 to 47, scores above 14 signifying severe bowel dysfunction.
Qualiveen questionnaire | At baseline, at 4 and 12 months; at 16 and 24 months
  Qualiveen questionnaire assesses neurogenic bladder function related quality of life, each item being scored on a Likert type scale ranging from 0 to 4, assessing 4 areas: discomfort, constraints, fears, and the patient's experience. The score ranges from 0 to 4, higher scores indicating lower bladder function related quality of life.
DN4 | At baseline, at 4 and 12 months; at 16 and 24 months
  DN4 questionnaire is used to identify neuropathic pain in patients. The score ranges from 0 to 10, a score of 4 or more is considered indicative of neuropathic pain.
Sensation assessment | At baseline, at 4 and 12 months; at 16 and 24 months
  3-item sensation assessment with binary choice responses (yes or no) assessed by a physician regarding participants' capacity to perceive superficial sensation (touch awareness, pain perception) and proprioceptive sensation (kinesthetic awareness).
Hospital Anxiety and Depression Scale | At baseline, at 4 and 12 months; at 16 and 24 months
  The Hospital Anxiety and Depression Scale is a 14-question instrument rated on a 4-point severity scale ranging between no impairment (0) and severe impairment (3). Hospital Anxiety and Depression Scale consists of two scales, one for anxiety, and one for depression, with a maximum score of 21 for each, respectively. Total scores from 8 to 10 for anxiety and depression are considered to be borderline abnormal and scores higher than 11 pathological.
Goal Attainment Scaling | At baseline, at 4 and 12 months; at 16 and 24 months
  Goal Attainment scaling tasks are individually identified to suit the subject, and the levels are individually set around their current and expected levels of performance. The progression is measured by identified levels that are as follows: Baseline score (-2), improved less than expected (-1), improved as expected (0), improved more than expected (+1) and improved much more than expected (+2).
The Sport Injury Rehabilitation Adherence Scale | At baseline, at 4 and 12 months; at 16 and 24 months
  The Sport Injury Rehabilitation Adherence Scale measures clinically-based adherence to rehabilitation. The overall score is 15, higher numbers, representing better adherence to rehabilitation.
Number of performed exoskeleton sessions | Weekly, up to 24 months for each participant
  The number of exoskeleton rehabilitation sessions performed will be tracked for each participant.
Duration of exoskeleton rehabilitation sessions | Weekly, up to 24 months for each participant
  The duration of exoskeleton rehabilitation sessions will be tracked for each participant, and will be expressed in minutes.
The duration of verticalization during exoskeleton rehabilitation sessions | Weekly, up to 24 months for each participant
  The time spent in an upright position (verticalization) during the exoskeleton rehabilitation sessions will be tracked for each participant, and expressed in minutes.
Number of steps performed during exoskeleton sessions | Weekly, up to 24 months for each participant
  The overall number of steps performed during the exoskeleton rehabilitation sessions will be tracked for each participant.
Level of device assistance during exoskeleton sessions | Weekly, up to 24 months for each participant
  The level of device assistance during the exoskeleton rehabilitation sessions will be tracked for each participant, and expressed as a percentage.
Number of passive steps performed during exoskeleton sessions | Weekly, up to 24 months for each participant
  The number of passive steps performed during the exoskeleton rehabilitation sessions will be tracked for each participant.
Number of active steps performed during exoskeleton sessions | Weekly, up to 24 months for each participant
  The number of active steps performed during the exoskeleton rehabilitation sessions will be tracked for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Sauvagnac, MD, Principal Investigator — Wandercraft
Locations (1):
- Wandercraft, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cieza A, Causey K, Kamenov K, Hanson SW, Chatterji S, Vos T. Global estimates of the need for rehabilitation based on the Global Burden of Disease study 2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2021 Dec 19;396(10267):2006-2017. doi: 10.1016/S0140-6736(20)32340-0. Epub 2020 Dec 1. PMID 33275908
- [Background] Eldar R, Kullmann L, Marincek C, Sekelj-Kauzlaric K, Svestkova O, Palat M. Rehabilitation medicine in countries of Central/Eastern Europe. Disabil Rehabil. 2008;30(2):134-41. doi: 10.1080/09638280701191776. PMID 17852214
- [Background] Kamenov K, Mills JA, Chatterji S, Cieza A. Needs and unmet needs for rehabilitation services: a scoping review. Disabil Rehabil. 2019 May;41(10):1227-1237. doi: 10.1080/09638288.2017.1422036. Epub 2018 Jan 5. PMID 29303004